CLINICAL TRIAL: NCT06301373
Title: Methotrexate Combined With Tofacitinib in the Treatment of Active Rheumatoid Arthritis With a Myeloid-stromal Pathotype: a Randomized, Controlled, Open Label, Multicenter Clinical Study
Brief Title: Methotrexate Combined With Tofacitinib in Rheumatoid Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-1185-02
Record Dates: First submitted 2024-01-22; First posted 2024-03-08 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Janus Kinase Inhibitors; Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate Combined With Tofacitinib (Experimental): Methotrexate 10-15mg orally once a week, tofacitinib 5mg orally twice a day
  Interventions: Drug: Methotrexate Combined With Tofacitinib
- Methotrexate (Active Comparator): Methotrexate 10-15mg orally once a week
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate Combined With Tofacitinib — Methotrexate Combined With Tofacitinib
  Other Names: JAK inhibitor
  Arms: Methotrexate Combined With Tofacitinib
Drug: Methotrexate — Methotrexate
  Arms: Methotrexate

SUMMARY:
Rheumatoid arthritis (RA) is the leading cause of disability in Chinese women. We established a synovial pathology queue in the early stage and proposed a new synovial immunopathology classification. We found that baseline myeloid stromal RA patients had severe conditions and poor outcome. Early identification of synovial myeloid stromal RA patients and intensified treatment are key to improving RA efficacy.

This project aims to conduct a randomized, controlled, open label, multicenter clinical study on early intensified treatment of RA based on synovial pathology classification. 130 adult patients with synovial myeloid stromal type of primary treatment moderate to severe active RA were planned to be enrolled in three centers: Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University; Shenshan Medical Center, Memorial Hospital of Sun Yat-Sen University, and Guangzhou Panyu Central Hospital. They were randomly divided into an intensive treatment group and a conventional treatment group in a 1:1 ratio. The intensive treatment group was treated with methotrexate combined with tofacitinib, while the conventional treatment group was treated with methotrexate monotherapy. The expected intervention period is 12 weeks, with a follow-up period of 48 weeks. The primary endpoint is the proportion of subjects who achieved ACR20 at week 12. Secondary endpoint indicators include improvement in disease activity and joint function among subjects at different follow-up points, safety, and the proportion of subjects who experienced joint destruction progression at week 48.

This project proposes the concept of achieving precise diagnosis of RA based on synovial pathology classification, and explores the efficacy of early methotrexate combined with tofacitinib intensified treatment for patients with synovial medullary stromal RA who have poor conventional treatment efficacy, providing high-level clinical evidence for achieving precise initial treatment of RA treatment guidelines.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is the leading cause of disability in Chinese women, but it cannot be cured. About 25%-40% of RA patients experience bone erosion within 6 months after experiencing joint symptoms. The first year after the onset of RA is the best window of treatment opportunity, and the earlier standardized treatment is initiated, the more effective RA treatment will be. RA patients have strong heterogeneity and lack effective evaluation indicators for early identification of patients with poor prognosis. Therefore, currently, domestic and foreign RA treatment guidelines do not include adverse prognostic factors in the initial stage. All RA patients are recommended to start treatment with methotrexate (MTX) monotherapy. If the improvement is not good after 3 months or does not meet the standard after 6 months, csDMARDs or targeted drug biologics or JAK inhibitors should be combined. However, clinical studies have found that the effective rate of MTX monotherapy after 3 months is only 30% to 50%, and most patients require combination therapy.

The pathological basis of RA is synovitis. In the early stage, we established a synovial pathology cohort and proposed a new synovial immunopathology classification. We found that baseline medullary stromal type (58%) RA patients had severe conditions, poor efficacy, and a risk of joint destruction progression after 1 year of imaging was 3.2 times higher than other types (Front Immunol, 2021), Among them, the efficacy of combining traditional synthetic DMARDs or biological agents for 3 months in the treatment of newly treated synovial medullary stromal RA patients is not as good as other types of patients [the core criteria for RA disease activity assessment of the American Society of Rheumatology reached 20% improvement (ACR20): 52% vs. 75%]. Therefore, early identification of patients with synovial myeloid stromal RA and intensified treatment are key to improving the efficacy of RA.

The plan for intensified treatment of RA includes the combination of MTX and biological agents or JAK inhibitors, where biological agents only target specific immune cells or cytokines, are expensive, require intravenous medication, and are prone to producing anti drug antibodies. JAK inhibitors can target JAK related inflammatory pathways in different cells, are convenient to take orally, and do not produce anti drug antibodies. The JAK inhibitors that have been listed in China include tofacitinib, Barretinib, and Upatinib. Among them, tofacitinib has the longest use time, good efficacy and safety, and is affordable after national centralized procurement, with strong promotability.

The characteristic of medullary stromal synovium is multicellular activation, which can secrete inflammatory factors and a large amount of matrix metalloproteinases (MMPs). It has been reported that tofacitinib can inhibit the production of synovial MMP-3. Our preliminary retrospective analysis showed that in RA patients with poor efficacy of csDMARDs or biologics, MTX combined with tofacitinib was used for treatment for 3 months, resulting in a 56% ACR20 and a significant decrease in serum MMP-3. This suggests that MTX combined with tofacitinib can be used as an intensive treatment for synovial myeloid stromal RA patients.

Based on this, we propose clinical questions: Synovial immunopathological classification helps to achieve accurate diagnosis of RA. Can MTX combined with tofacitinib intensive treatment be applied to newly treated RA patients with synovial myeloid stromal type to achieve early disease control?

This project aims to conduct a randomized, controlled, open label, multicenter clinical study on early intensified treatment of RA based on synovial pathology classification. 130 newly treated adult patients with moderate to severe active rheumatoid arthritis (RA) of the synovial medullary matrix type were randomly divided into an intensive treatment group and a conventional treatment group in a 1:1 ratio. The intensive treatment group was treated with MTX combined with tofacitinib, while the conventional treatment group was treated with MTX monotherapy. The expected intervention period is 12 weeks, with a follow-up period of 48 weeks. The primary endpoint is the proportion of subjects who achieved ACR20 at week 12. Secondary endpoint indicators include improvement in disease activity and joint function among subjects at different follow-up points, safety, and the proportion of subjects who experienced joint destruction progression at week 48. The exploratory objective (sub topic) is to apply proteomics to screen serum biomarkers in patients with synovial myeloid stromal RA and establish a precise diagnostic system.

This project is based on the applicant's long-term research on synovial pathology of RA, proposing the concept of achieving accurate diagnosis of RA based on synovial pathology classification. At the same time, it aims to explore the efficacy of early MTX combined with tofacitinib in patients with synovial medullary stromal RA who have poor conventional treatment efficacy, providing high-level clinical evidence for achieving precise initial treatment of RA treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed according to the 1987 American College of Rheumatology or 2010 American College of Rheumatology/European League Against Rheumatism criteria
* Patients had moderate or high disease activity
* Patients had a synovial biopsy and with a myeloid-stromal pathotype
* Patients with good compliance, willing to participate in this study and sign an informed consent form

Exclusion Criteria:

* Patient received conventional synthetic disease modifying anti-rheumatic drugs treatment in the first 12 weeks of randomization
* Patient received biologic agents treatment in the first 6 months of randomization
* Patient received Janus kinase inhibitor treatment before randomization
* Patient with serious diseases under control (such as diabetes), serious respiratory diseases, serious chronic gastrointestinal diseases (such as active or recurrent gastrointestinal ulcers), serious blood system diseases (such as aplastic anemia, myelodysplastic syndrome) or any disease that can cause hemolysis or erythrocyte instability (such as malaria, hemolytic anemia)
* Patients with moderate to severe congestive heart failure (New York Heart Association grade III or IV), or recent (within 6 months prior to screening) cerebrovascular accident, myocardial infarction, coronary stent implantation, or uncontrolled hypertension
* Patients with blood routine WBC<4.0 × 109/L, and/or Hb<90g/L, and/or Plt<100 × 109/L during the screening period
* Patients with active chronic liver disease or abnormal liver function, AST, ALT, GGT, and TBIL are more than twice the upper limit of normal during the screening period
* Patients with estimated glomerular filtration rate <30ml/min during screening period
* Patients with history of symptomatic herpes zoster infection (within the first 12 weeks of randomization), recurrent or disseminated (even if only once) herpes zoster or disseminated (even if only once) herpes simplex infection
* Chest X-ray or CT examination indicates active tuberculosis, or latent tuberculosis (T-SPOT or TB-IGRA positive) without prophylactic tuberculosis treatment for at least 4 weeks
* Patients woth hepatitis C virus ribonucleic acid (HCV-RNA) testing are higher than the lower limit of detection; Or positive for Treponema pallidum antibody (TP Ab); Or human immunodeficiency virus antibody (HIV Ab) positive during the selected period
* Patients with hepatitis B surface antigen positive without prophylactic antiviral treatment
* Patients with history of lymphoproliferative diseases, or possibly various signs or symptoms of lymphoproliferative diseases
* Patients with any active malignant tumors or history of malignant tumors within the first 5 years, except for skin squamous or basal cell carcinoma, cervical carcinoma in situ, or breast ductal carcinoma in situ that has been treated and considered cured
* Patients with history of thromboembolism, including deep vein thrombosis, pulmonary embolism, arterial thrombosis, etc., or high risk factors prone to thromboembolism (such as obesity, smoking, abnormal coagulation function, diabetes, long-term use of estrogen or use of compound hormonal contraceptives or hormone replacement therapy, long-term braking, etc., which are comprehensively judged by the investigator according to clinical evaluation)
* Patients with undergone major surgery within the first 4 weeks of randomization, or is expected to undergo major surgery after enrollment; Or a history of chronic pain that may affect the evaluation of the study; Or have received organ transplantation before
* Patients with history of mental illness, alcoholism, drug or other substance abuse
* Pregnant women, lactating women, and men or women who plan to conceive in the near future
* The researchers believe that there are any other factors that may affect the progress or evaluation of the results of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who achieved ACR20 | 12 week
  ACR20

SECONDARY OUTCOMES:
Changes in disease activity scores (DAS28-CRP) relative to baseline | 4, 8, 12, 24, 36, and 48 weeks after treatment
  DAS28-CRP
Changes in disease activity scores (DAS28-ESR) relative to baseline | 4, 8, 12, 24, 36, and 48 weeks after treatment
  DAS28-ESR
Changes in disease activity scores (SDAI) relative to baseline | 4, 8, 12, 24, 36, and 48 weeks after treatment
  SDAI
Changes in disease activity scores (CDAI) relative to baseline | 4, 8, 12, 24, 36, and 48 weeks after treatment
  CDAI
Proportion of subjects with low disease activity and remission (SDAI standard) at weeks 4, 8, 12, 24, 36, and 48 after treatment | 4, 8, 12, 24, 36, and 48 weeks after treatment
  low disease activity and remission
The proportion of subjects who met ACR50 criteria at weeks 4, 8, 12, 24, 36, and 48 after treatment | 4, 8, 12, 24, 36, and 48 weeks after treatment
  ACR50
The proportion of subjects who met ACR70 criteria at weeks 4, 8, 12, 24, 36, and 48 after treatment | 4, 8, 12, 24, 36, and 48 weeks after treatment
  ACR70
Changes in the Disability Index (HAQ-DI) of the Health Assessment Questionnaire relative to baseline | 4, 8, 12, 24, 36, and 48 weeks after treatment
  HAQ-DI
Changes in EQ-5D-5L relative to baseline | 4, 8, 12, 24, 36, and 48 weeks after treatment
  EQ-5D-5L
The proportion of subjects with joint destruction progression at 48 weeks after treatment | 48 weeks
  joint destruction progression

OTHER OUTCOMES:
The proportion of adverse events (AE) in subjects at 4, 8, 12, 24, 36, and 48 weeks after treatment | 4, 8, 12, 24, 36, and 48 weeks after treatment
  adverse events (AE)
The proportion of severe adverse events (SAE) in subjects at 4, 8, 12, 24, 36, and 48 weeks after treatment | 4, 8, 12, 24, 36, and 48 weeks after treatment
  severe adverse events (SAE)
Changes in serum MMP-3 levels relative to baseline | 4, 8, 12, 24, 36, and 48 weeks after treatment
  serum MMP-3 levels

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China